CLINICAL TRIAL: NCT07346807
Title: A Phase II Single-Arm Study of Lingual Nerve Disruption to Augment Neoadjuvant Chemoimmunotherapy in Locally Advanced Tongue Cancer
Brief Title: Lingual Nerve Disruption to Augment Neoadjuvant Chemoimmunotherapy in Locally Advanced Tongue Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-792R
Record Dates: First submitted 2025-12-24; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Tongue Squamous Cell Carcinoma
MeSH Terms: interventions — tislelizumab; Albumin-Bound Paclitaxel; Cisplatin; Monitoring, Immunologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lingual Nerve Disruption + Neoadjuvant Chemoimmunotherapy (Experimental)
  Interventions: Procedure: Lingual Nerve Disruption; Drug: Tislelizumab; Drug: Albumin-bound Paclitaxel; Procedure: Cisplatin; Procedure: Peripheral Blood Collection for Immune Monitoring; Other: Pain and Quality of Life Assessment

INTERVENTIONS:
Procedure: Lingual Nerve Disruption — Surgical transection of 1 cm of the lingual nerve via intraoral approach under local anesthesia at the time of biopsy. This procedure induces ipsilateral tongue tip numbness to enhance subsequent chemoimmunotherapy efficacy.
Drug: Tislelizumab — Anti-PD-1 monoclonal antibody administered intravenously at 200 mg on day 1 of each 3-week cycle.
Drug: Albumin-bound Paclitaxel — Chemotherapy agent administered intravenously at 260 mg/m² on day 2 of each 3-week cycle.
Procedure: Cisplatin — Chemotherapy agent administered intravenously at 75 mg/m² on day 2-3 of each 3-week cycle.
Procedure: Peripheral Blood Collection for Immune Monitoring — Peripheral blood (10 mL) collected in the morning under fasting conditions at baseline, before each cycle of neoadjuvant therapy, and during follow-up visits. Plasma and peripheral blood mononuclear cells are prepared within 2 hours and stored at -80°C for immune cell dynamic analysis.
Other: Pain and Quality of Life Assessment — McGill Pain Questionnaire and quality-of-life surveys administered before each cycle of neoadjuvant therapy to assess treatment impact on pain relief and functional outcomes.

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility and preliminary efficacy of lingual nerve disruption combined with neoadjuvant chemoimmunotherapy in patients with locally advanced tongue squamous cell carcinoma.

The study aims to learn whether surgical disruption of the lingual nerve can enhance the effectiveness of neoadjuvant chemoimmunotherapy before definitive surgery in adults with locally advanced (cT3/T4) tongue cancer. The main questions it aims to answer are:

Can lingual nerve disruption combined with neoadjuvant chemoimmunotherapy improve tumor response prior to surgery?

Is this combined treatment approach safe and feasible for patients with locally advanced tongue cancer?

This is a single-arm, phase II clinical trial.

Participants will:

Undergo tumor biopsy with simultaneous surgical disruption of the affected-side lingual nerve.

Receive neoadjuvant chemoimmunotherapy consisting of tislelizumab, cisplatin, and nab-paclitaxel for two treatment cycles.

Undergo definitive surgical resection of the primary tumor and neck dissection.

Attend scheduled follow-up visits for safety assessments, imaging evaluations, and collection of blood samples for immune monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years, male or female.
2. Histologically or cytologically confirmed primary tongue squamous cell carcinoma (cT3 or cT4).
3. Patients scheduled to receive 2 cycles of preoperative neoadjuvant chemoimmunotherapy with tirelizumab, cisplatin, and albumin-bound paclitaxel.
4. Patients planned to undergo surgical resection of tongue cancer following neoadjuvant therapy.
5. Voluntary participation with signed informed consent, good compliance, and willingness to follow study procedures.

Exclusion Criteria:

1. Known distant metastases of the tumor.
2. History of tongue squamous cell carcinoma or other malignant tumors of the tongue within the past 5 years.
3. Active infection requiring systemic therapy; non-infectious pneumonia or interstitial lung disease requiring steroid therapy, or current pneumonia/interstitial lung disease; known hepatitis B infection (HBsAg positive) or active hepatitis C infection (detectable HCV RNA); known HIV infection.
4. Previous allogeneic tissue or organ transplantation.
5. Unresolved ≥Grade 2 (CTCAE v5.0) toxicities from prior anticancer treatments, except alopecia.
6. Significant cardiovascular abnormalities (e.g., myocardial infarction, superior vena cava syndrome, NYHA class ≥II heart disease within 3 months prior to enrollment).
7. Active serious clinical infections (>Grade 2 NCI-CTCAE v5.0).
8. Uncontrolled hypertension (treated systolic BP >150 mmHg and/or diastolic BP >90 mmHg) or clinically significant cardiovascular disease, including recent cerebrovascular accident or myocardial infarction (≤6 months), unstable angina, NYHA class ≥II congestive heart failure, or severe arrhythmia not controlled by medication that could affect study treatment.
9. Laboratory abnormalities:

   Hematology: WBC <3,000/mm³, Hb <8 g/dL, platelets <80,000/mm³ Liver function: ALT/AST >3× upper limit of normal, bilirubin >1.5× ULN Renal function: serum creatinine >1.5× ULN, renal failure requiring dialysis Diabetes: poorly controlled (FBG >10 mmol/L) Proteinuria: urine protein ≥++ and 24-hour urine protein >1.0 g
10. Pregnant women; breastfeeding women must discontinue breastfeeding to participate.
11. History of substance abuse or psychiatric disorders that would interfere with study participation.
12. Participation in another clinical trial within 30 days prior to enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Major Pathologic Response (MPR) Rate | From baseline (day1, before biopsy and lingual nerve disruption) to surgery (3 weeks after completion of 2 cycles of neoadjuvant therapy, which starts 1 week after the biopsy. Each cycle of neoadjuvant therapy is 21 days/3 weeks)

SECONDARY OUTCOMES:
Preoperative Pain Score Improvement Rate | From baseline (day1, before biopsy and lingual nerve disruption) to surgery (3 weeks after completion of 2 cycles of neoadjuvant therapy, which starts 1 week after the biopsy. Each cycle of neoadjuvant therapy is 21 days/3 weeks)

OTHER OUTCOMES:
Dynamic Changes of Immune Cells | At 5 specific time points during the study: Baseline (day1) Before second cycle of neoadjuvant therapy (day28 / 4 weeks) After second cycle of neoadjuvant therapy before surgery (day49 / 7weeks) 4 weeks after surgery(day77) 3 months after surgery(day139)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No